CLINICAL TRIAL: NCT02719912
Title: Mitral Valve Replacement With the MValve Dock and A Percutaneous Transcatheter Heart Valve
Brief Title: Mitral Valve Replacement With MValve Dock and Lotus
Acronym: DOCK 1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: MValve Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP 01-2015
Record Dates: First submitted 2016-03-21; First posted 2016-03-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Mitral Valve Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Valve Replacement (Experimental): Mitral valve replacement
  Interventions: Device: mitral valve replacement

INTERVENTIONS:
Device: mitral valve replacement — transcatheter mitral valve replacement

SUMMARY:
This study evaluates the MValve mitral prosthesis in conjunction with a Lotus transcatheter heart valve (THV) for mitral valve replacement in subjects at high risk for conventional mitral valve replacement or repair surgery.

DETAILED DESCRIPTION:
This study is a prospective first in man feasibility study intended to evaluate preliminary safety and effectiveness of the MValve Mitral Dock with Lotus transcatheter heart valve for mitral valve replacement in subjects who are at high risk for surgical valve repair or replacement.

The surgical technique adapts the valve-in-valve approach for mitral replacement in degenerated mitral prostheses to failing native mitral valves. The MValve Dock is designed to provide a structural platform within the mitral annulus so that the Lotus THV can be implanted in a secure fashion in the mitral annulus. The investigational device anchors to the mitral annulus commissures, sparing the native valve leaflets and sub annular apparatus. This study is designed to treat subjects with moderate-to-severe MR who are not deemed candidates for mitral valve surgery.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic ≥3+ degenerative or functional mitral regurgitation of either ischemic or non-ischemic etiology based by a qualifying echocardiography obtained within 90 days prior to the procedure.
* New York Heart Association (NYHA) Functional Class III or IV.
* High risk for conventional open mitral valve repair or replacement surgery in the consideration of the site Heart Team.
* Left Ventricular Ejection Fraction (LVEF) is ≥30% within 30 days prior to the procedure.
* Mitral valve annular commissure to commissure (C/C) dimension between 30-35 mm by echocardiography.
* Left atrial diameter <5.5 cm by echocardiography

Exclusion Criteria:

* Prior mitral valve replacement or repair surgery.
* Prior transapical surgery.
* Severe aortic or tricuspid valve disease. - Severe symptomatic carotid stenosis (>70% by ultrasound).
* ACC/AHA Stage D heart failure.
* Hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, or any other structural heart disease causing heart failure other than dilated cardiomyopathy of either ischemic or non-ischemic etiology.
* Infiltrative cardiomyopathies (amyloidosis, hemochromatosis, sarcoidosis).
* Physical evidence of right-sided congestive heart failure with echocardiographic evidence of moderate or severe right ventricular dysfunction.
* Severe mitral annular calcification.
* Glomerular filtration rate (GFR) < 30.
* Hemodynamic instability defined as systolic pressure < 90 mm Hg with or without afterload reduction, cardiogenic shock, or the need for inotropic support or intra-aortic balloon pump or other hemodynamic support device, or any mechanical heart assistance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Composite serious adverse cardiac events and stroke | 30 days
  death, myocardial infarction, stroke, repeat surgery

SECONDARY OUTCOMES:
Mitral regurgitation grade | 1 year

CONTACTS AND LOCATIONS:
Locations (4):
- Dante Pazzenese Institute of Cardiology, Sau Paulo, Brazil
- Clinique Pasteur, Toulouse, France
- University of Bonn - Medizinische Klinik und Poliklinik II, Bonn, Germany
- University of Poznan, Poznan, Poland